CLINICAL TRIAL: NCT03629041
Title: A Study of the Use of Microneedle Patches to Deliver Topical Lidocaine in the Oral Cavity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innoture Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Innoture/NW-01
Record Dates: First submitted 2018-07-24; First posted 2018-08-14 (Actual); Results first posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-10

CONDITIONS: Topical Anaesthesia
MeSH Terms: interventions — Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment A - Microneedle patch (Experimental): The application of a 5% topical lidocaine gel to one of the identified areas within the participants mouth using a microneedle patch. The microneedle patch will be applied to the oral mucosa of the identified site for 3 minutes, followed by infiltration with local anaesthetic to one of the identified areas within the participants mouth.
  Interventions: Device: Microneedle Patch
- Treatment B - Patch with no microneedles (Sham Comparator): The application of a 5% topical lidocaine gel to one of the identified sites within the participants mouth using a patch with no microneedles. The patch with no microneedles will be applied to the oral mucosa of the identified site for 3 minutes, followed by infiltration with local anaesthetic to one of the identified areas within the participants mouth.
  Interventions: Device: Patch with no microneedles

INTERVENTIONS:
Device: Microneedle Patch — At the first visit participants will have either the buccal or palatal treated. At the second visit the other area will be treated.
  Arms: Treatment A - Microneedle patch
Device: Patch with no microneedles — At the first visit participants will have either the buccal or palatal treated. At the second visit the other area will be treated.
  Arms: Treatment B - Patch with no microneedles

SUMMARY:
To look at the effect on patient perceived pain resulting from infiltration injection with local anaesthetic in a dental syringe with prior application of topical anaesthetic to the oral mucosa on a microneedle patch compared to a patch with no microneedles. To look at the safety of the patches when applied to the oral mucosa.

DETAILED DESCRIPTION:
This is a randomised, 2 treatment, double blind design, with respect to the clinical assessor and subject, split mouth, crossover design with a negative control (patch with no microneedles).

Potential participants will be invited to attend a screening visit. At this visit participants will be asked to read and sign a Participant Information Sheet and Consent Form prior to any study procedures being performed. They will be given ample time to decide if they wish to participate in the study.

A dentally qualified clinician will record the participant's demographics, medical history, current/concomitant medications, perform an oral soft tissue examination and ensure the participant fulfils the inclusion and exclusion criteria for the study. Two areas of the mouth will be identified for assessment during the study. The areas of the mouth will be identified as S1 or S2. Site S1 will be left or right palatal mucosa adjacent to the premolar area and S2 will be left or right upper buccal mucosa adjacent to the upper lateral incisor area.

Participants who successfully fulfil all the necessary entrance criteria will be provided with training by study staff on how to use a VAS record sheet and randomised on to the study to receive treatment combination A or B at in a random order according to a predetermined randomisation schedule supplied by the study statistician. The screening visit and first treatment visit will occur at the same visit. The treatment possibilities are outlined below:

Treatment A The application of a 5% topical lidocaine gel to one of the identified areas within the participants mouth using a microneedle patch. The microneedle patch will be applied to the oral mucosa of the identified site for 3 minutes, followed by infiltration with local anaesthetic to one of the identified areas within the participants mouth.

Treatment B The application of a 5% topical lidocaine gel to one of the identified sites within the participants mouth using a patch with no microneedles. The patch with no microneedles will be applied to the oral mucosa of the identified site for 3 minutes, followed by infiltration with local anaesthetic to one of the identified areas within the participants mouth.

The chosen sites will be: S1; left and right palatal mucosa adjacent to the premolar area or S2; left and right upper buccal mucosa adjacent to the upper lateral incisor area. Each participant at the first visit will have either S1 or S2 sites allocated for treatment. For example, Treatment A will be allocated to S1 left side and Treatment B to S1 right side or vice versa. At the second visit, 2 weeks (+/- 3 days) after the first visit, Treatment B will be allocated to S2 left side and Treatment A to S2 right side. Both sides of the mouth for S1 or S2 will be treated at the same. After each treatment participants will be asked to make pain assessments relating to needle insertion into the oral mucosa and the giving of the local infiltration anaesthetic.

It is envisaged that a sufficient number of potential participants will be screened in order to randomise 16 onto the study.

Assessment methods: Pain assessments will be performed after application of the topical anaesthetic for 3 minutes. Each test will be performed sequentially i.e. 3 separate needle insertions, with pain assessments recorded by the participant using a Visual Analogue Scale (VAS) and a verbal pain grading after each test. The level of pain at S1 or S2 will be assessed as follows:

Test I. A short dental needle, mounted on a dental syringe containing a cartridge of 2% lidocaine hydrochloride and 1:80,000 adrenaline, will be used to penetrate the oral mucosa at the treated site and the patient asked to score the pain using a VAS rating scale and by verbal grading of zero, mild, moderate or severe.

Test 2. The same needle will be inserted through the oral mucosa and down to contact bone. Pain will be assessed as in Test 1.

Test 3. The same needle will be again inserted through the oral mucosa and the cartridge of local anaesthetic will be injected into the site. Pain will be again assessed as in Test I.

Following enrolment on to the study, participants will be given written and verbal instructions on the VAS and how to complete it.

ELIGIBILITY:
Inclusion Criteria:

1. be aged 18 years and over, of either gender and in good health;
2. be willing and physically able to carry out all study procedures;
3. be willing and able to give Informed Consent and provide details of any medical history;
4. be available for all of the study dates
5. have a good standard of oral hygiene and gingival health
6. must have 1 premolar or canine in each quadrant that has no/minimal restorations

Exclusion Criteria:

1. presence of soft tissue oral pathology;
2. presence of advanced periodontal disease;
3. Individuals with any serious health conditions, that would preclude participation, in the professional judgement of the Study Dentist;
4. individuals with known allergies or sensitivities to local anaesthetics
5. have participated in another clinical trial in the last 30 days
6. in the opinion of the investigator unable to comply fully with the trial requirements.
7. the subject is an employee of the Sponsor or the site conducting the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicola X West, Principal Investigator — Bristol Dental School
Locations (1):
- Rhiwbina Dental Surgery, Cardiff, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were healthy volunteers who have their regular dental care at Rhiwbina Dental Surgery.
Groups:
- Treatment Group 1: At visit 1 the left upper palatal area was treated with lidocaine on a microneedle patch for three minutes and the right upper palatal area was treated with lidocaine on a patch with no microneedles for three minutes. Tests 1, 2 and 3 were then performed on both sites.
  At visit 2 (2 weeks +/- 3 days after visit 1) the left upper anterior buccal sulcus was treated with lidocaine on a patch with no microneedles for three minutes and the right upper anterior buccal sulcus was treated with lidocaine on a microneedle patch for three minutes. Tests 1, 2 and 3 were then performed on both sites.
- Treatment Group 2: At visit 1 the left upper palatal area was treated with lidocaine on a patch with no microneedles for three minutes and the right upper palatal area was treated with lidocaine on a microneedle patch for three minutes. Tests 1, 2 and 3 were then performed on both sites.
  At visit 2 (2 weeks +/- 3 days from visit 1) the left upper anterior buccal sulcus was treated with lidocaine on a microneedle patch for three minutes and the right upper anterior buccal sulcus was treated with lidocaine on a patch with no microneedles for three minutes. Tests 1, 2 and 3 were then performed on both sites.
- Treatment Group 3: At visit 1 the left upper anterior buccal sulcus was treated with lidocaine on a microneedle patch for three minutes and the right upper anterior buccal sulcus was treated with lidocaine on a patch with no microneedles for three minutes. Tests 1, 2 and 3 were then performed on both sites.
  At visit 2 (2 weeks +/- 3 days from visit 1) the left upper palatal area was treated with lidocaine on a patch with no microneedles for three minutes and the right upper palatal area was treated with lidocaine on a microneedle patch for three minutes. Tests 1, 2 and 3 were then performed on both sites.
- Treatment Group 4: At visit 1 the left upper anterior buccal sulcus was treated with lidocaine on a patch with no microneedles for three minutes and the right upper anterior buccal sulcus was treated with lidocaine on a microneedle patch for three minutes. Tests 1, 2 and 3 were then performed on both sites.
  At visit 2 (2 weeks +/- 3 days after visit 1) the left upper palatal area was treated with lidocaine on a microneedle patch for three minutes and the right upper palatal area was treated with lidocaine on a patch with no microneedles for three minutes. Tests 1, 2 and 3 were then performed on both sites.
Period: Visit 1
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Visit 2 (2 Weeks ± 3 Days From Visit 1)
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4
Started | 4 | 4 | 4 | 4
Completed | 4 | 3 | 4 | 4
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 31.4 [18.9 to 57.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 16

OUTCOME MEASURES:

1. Primary Outcome: VAS in Healthy Participants, When Topical 5% Lidocaine Dental Gel Was Applied to the Upper Palatal and Upper Anterior Buccal Sulcus Areas With a Microneedle Patch and a Patch With no Microneedles, Prior to Infiltration With Local Anaesthesia.
Description: Pain levels were recorded using a visual analogue scale (VAS). When responding to the VAS item, subjects were required to indicate their level of pain by indicating a position along a continuous line between two end-points of no pain (0) and worst pain imaginable (100). The lower the score the better the outcome. The topical lidocaine was applied either with a microneedle patch or a patch with no microneedles for 3 minutes. Immediately afterwards three tests were performed: Test 1, a short dental needle, mounted on a dental syringe containing a cartridge of 2% lidocaine hydrochloride and 1:80,000 adrenaline, was used to penetrate the oral mucosa at the treated site; test 2, the same needle was inserted through the oral mucosa and down to contact bone; test 3, the same needle was again inserted through the oral mucosa and the cartridge of local anaesthetic was injected into the site.
Time Frame: Following 3 minutes of application of topical anaesthetic using a patch, the 3 tests were performed and the pain score recorded immediately after each test.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment A - Microneedle Patch, Palatal: The application of a 5% topical lidocaine gel to the palatal mucosa within the participants mouth using a microneedle patch. The microneedle patch was applied to the palatal mucosa for 3 minutes, followed by infiltration with local anaesthetic to the palatal mucosa within the participants mouth.
- Treatment B - Patch With no Microneedles, Palatal: The application of a 5% topical lidocaine gel to the palatal mucosa sites within the participants mouth using a patch with no microneedles. The patch with no microneedles was applied to the palatal mucosa for 3 minutes, followed by infiltration with local anaesthetic to the palatal mucosa within the participants mouth.
- Treatment A - Microneedle Patch, Buccal: The application of a 5% topical lidocaine gel to the buccal mucosa within the participants mouth using a microneedle patch. The microneedle patch was applied to the buccal mucosa for 3 minutes, followed by infiltration with local anaesthetic to the buccal mucosa within the participants mouth.
- Treatment B - Patch With no Microneedles, Buccal: The application of a 5% topical lidocaine gel to the buccal mucosa sites within the participants mouth using a patch with no microneedles. The patch with no microneedles was applied to the buccal mucosa for 3 minutes, followed by infiltration with local anaesthetic to the buccal mucosa within the participants mouth.
Arm/Group | Treatment A - Microneedle Patch, Palatal | Treatment B - Patch With no Microneedles, Palatal | Treatment A - Microneedle Patch, Buccal | Treatment B - Patch With no Microneedles, Buccal
Number analyzed (Participants) | 16 | 16 | 15 | 15
units on a scale
  VAS scores, test 1 | 5.1 (5.8) | 12.3 (11.6) | 0.7 (1.0) | 4.0 (5.8)
  VAS scores, test 2 | 11.9 (11.3) | 18.7 (12.4) | 2.8 (4.0) | 6.9 (6.6)
  VAS scores, test 3 | 26.8 (20.1) | 39.5 (25.1) | 18.3 (17.5) | 30.6 (20.7)

2. Primary Outcome: Verbal Pain Grading, When Topical 5% Lidocaine Dental Gel is Applied to the Upper Palatal and Upper Anterior Buccal Sulcus Areas With a Microneedle Patch and a Patch With No Microneedle Patch, Prior to Infiltration With Local Anaesthesia. Test 1
Description: Pain levels will be recorded using a Verbal Pain Grading. For the verbal pain grading, subjects are asked to score either zero, mild, moderate or severe. In test 1, a short dental needle, mounted on a dental syringe containing a cartridge of 2% lidocaine hydrochloride and 1:80,000 adrenaline, was used to penetrate the oral mucosa at the treated site.
Time Frame: Following three minutes of application of topical anaesthetic with a patch, the 3 tests were performed and the pain score recorded immediately after each test.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment A - Microneedle Patch, Palatal: 5% topical lidocaine gel was applied to the upper palatal area within the participants mouth using a microneedle patch. The microneedle patch was applied for 3 minutes and then removed, followed by tests 1, 2 and 3.
- Treatment B - Patch With no Microneedles, Palatal: 5% topical lidocaine gel was applied to the upper palatal area within the participants mouth using a patch with no microneedles. The patch with no microneedles was applied for 3 minutes and then removed, followed by tests 1, 2 and 3.
- Treatment A - Microneedle Patch, Buccal: 5% topical lidocaine gel was applied to the upper anterior buccal sulcus within the participants mouth using a microneedle patch. The microneedle patch was applied for 3 minutes and then removed, followed by tests 1, 2 and 3.
- Treatment B - Patch With no Microneedles, Buccal: 5% topical lidocaine gel was applied to the upper anterior buccal sulcus within the participants mouth using a patch with no microneedles. The patch with no microneedles was applied for 3 minutes and then removed, followed by tests 1, 2 and 3.
Arm/Group | Treatment A - Microneedle Patch, Palatal | Treatment B - Patch With no Microneedles, Palatal | Treatment A - Microneedle Patch, Buccal | Treatment B - Patch With no Microneedles, Buccal
Number analyzed (Participants) | 16 | 16 | 15 | 15
Participants
  Verbal Pain Grading, Test 1- Zero | 8 | 5 | 15 | 13
  Verbal Pain Grading, Test 1 - Mild | 8 | 8 | 0 | 2
  Verbal Pain Grading, Test 1 - Moderate | 0 | 3 | 0 | 0
  Verbal Pain Grading, Test 1 - Severe | 0 | 0 | 0 | 0

3. Secondary Outcome: Adverse Events in Healthy Participants When a Proprietary Topical 5% Lidocaine Dental Gel Was Applied to the Oral Mucosa With a Microneedle Patch and a Patch With no Microneedles, Prior to Infiltration With Local Anaesthesia.
Description: Adverse events were recorded
Time Frame: Events were collected from the time of informed consent until end of treatment or when an ongoing AE had resolved whichever was latest, unless the PI & the Innoture contact from the clinical investigation plan agreed that no further follow up was needed.
Measure: Number; unit: Events
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4
Number analyzed (Participants) | 4 | 4 | 4 | 4
Events | 0 | 0 | 0 | 0

4. Primary Outcome: Verbal Pain Grading, When Topical 5% Lidocaine Dental Gel Was Applied to the Upper Palatal and Upper Anterior Buccal Sulcus Areas With a Microneedle Patch and a Patch With No Microneedle Patch, Prior to Infiltration With Local Anaesthesia. Test 2
Description: Pain levels were recorded using a Verbal Pain Grading. For the verbal pain grading, subjects were asked to score either zero, mild, moderate or severe. In test 2, the same needle as test 1 was inserted through the oral mucosa and down to contact bone.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A - Microneedle Patch, Palatal | Treatment B - Patch With no Microneedles, Palatal | Treatment A - Microneedle Patch, Buccal | Treatment B - Patch With no Microneedles, Buccal
Number analyzed (Participants) | 16 | 16 | 15 | 15
Participants
  Verbal Pain Grading, Test 2 - Zero | 8 | 3 | 14 | 11
  Verbal Pain Grading, Test 2 - Mild | 5 | 9 | 1 | 4
  Verbal Pain Grading, Test 2 - Moderate | 3 | 4 | 0 | 0
  Verbal Pain Grading, Test 2 - Severe | 0 | 0 | 0 | 0

5. Primary Outcome: Verbal Pain Grading, When Topical 5% Lidocaine Dental Gel Was Applied to the Upper Palatal and Upper Anterior Buccal Sulcus Areas With a Microneedle Patch and a Patch With No Microneedle Patch, Prior to Infiltration With Local Anaesthesia. Test 3
Description: Pain levels were recorded using a Verbal Pain Grading. For the verbal pain grading, subjects were asked to score either zero, mild, moderate or severe. In test 3, the same needle as test 1 and test 2 was again inserted through the oral mucosa and the cartridge of local anaesthetic was injected into the site.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A - Microneedle Patch, Palatal | Treatment B - Patch With no Microneedles, Palatal | Treatment A - Microneedle Patch, Buccal | Treatment B - Patch With no Microneedles, Buccal
Number analyzed (Participants) | 16 | 16 | 15 | 15
Participants
  Verbal Pain Grading, Test 3 - Zero | 1 | 1 | 3 | 1
  Verbal Pain Grading, Test 3 - Mild | 7 | 3 | 8 | 7
  Verbal Pain Grading, Test 3 - Moderate | 8 | 10 | 4 | 7
  Verbal Pain Grading, Test 3 - Severe | 0 | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent until end of treatment or when an ongoing AE had resolved whichever was latest, unless the PI and the Innoture contact named in the clinical investigation plan agreed that no further follow up was necessary.
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT03629041/Prot_SAP_000.pdf